CLINICAL TRIAL: NCT04379362
Title: Magnetic Resonance Imaging-guided Focal Laser Ablation of Prostate Cancer
Brief Title: MRI-guided Focal Laser Ablation
Acronym: Unicorn
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Biolitec (Unknown); Soteria Medical (Unknown); Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL63647.091.17
Record Dates: First submitted 2020-04-23; First posted 2020-05-07 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer
Keywords: Focal laser ablation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-center, interventional treatment, non-randomized, open label, single arm, phase II study with a medical device.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low or intermediate grade prostate cancer (Experimental)
  Interventions: Procedure: Focal laser ablation

INTERVENTIONS:
Procedure: Focal laser ablation — Focal laser ablation

SUMMARY:
Magnetic resonance imaging-guided focal laser ablation of prostate cancer.

ELIGIBILITY:
Inclusion criteria:

* MRI visible index lesion (on T2-weighted MR imaging or diffusion weighted imaging);
* Maximum MRI visible lesion size is ≤ 15 mm large axis;
* Life expectancy at inclusion of more 10 years;
* Diagnosis of prostate cancer confirmed by targeted biopsy using TRUS-MRI fusion or in-bore MRI guided biopsies;
* Criteria of low and intermediate risk of progression and eligibility for focal therapy (clinical stage of maximum T2c, maximum biopsy Gleason score of 4 + 3 on targeted biopsies, serum prostate specific antigen < 15 ng/ml);
* Patient accepting to be included in an active surveillance protocol at the end of the study, in accordance with the recommendations of good practice.

Exclusion criteria:

* History of prostate surgery;
* History of radiation therapy or pelvic trauma; history of proved acute or chronic prostatitis;
* History of tumor in the preceding 5 years (excluded: non-metastatic basal cell skin cancer);
* Severe urinary symptoms associated with benign hyperplasia of the prostate, and defined by an IPSS score > 18;
* Tumor with MRI signs of extra-capsular extension or invasion of the seminal vesicles;
* Maximum cancer core length >3 mm and/or maximum Gleason score of 3+4 on systematic biopsies outside the visible tumor area on mpMRI;
* Impossibility to obtain a valid informed consent;
* Patients unable to undergo MR imaging, including those with contra-indications;
* Contra-indications to MR guided focal laser therapy (colitis ulcerosa, rectal pathology or abdomino perineal resection);
* Metallic hip implant or any other metallic implant or device that distorts local magnetic field and compromises the quality of MR imaging;
* Patients with evidence for nodal or metastatic disease;
* Patients with an estimated Glomerular Filtration Ratio (eGFR) < 40 mL/min/1.73 m2.

Ages: 45 Years to 76 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender identity
Enrollment: 53 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Urine incontinence incontinence | At inclusion, 3 months, 6 months, 12 months and 24 months follow up.
  To evaluate a change in the functional outcome urine incontinence before and after FLA in patients with localized low to intermediate risk prostate cancer (Gleason 3+3, 3+4 or Gleason 4+3).

SECONDARY OUTCOMES:
Local cancer control | At inclusion , 3 months, 6 months, 12 months and 24 months follow up.
  To assess the safety outcome local cancer control achieved at the ablation site after FLA by multiparametric MR imaging and targeted prostate biopsies.
International Prostate Symptom Score (IPSS) | At inclusion, 3 months, 6 months, 12 months and 24 months follow up.
  To evaluate other functional outcomes (sexual, hormonal and bowel functions) before and after FLA in men with prostate cancer by using validated questionnaires e.g. International Prostate Symptom Score (IPSS)
Sexual Health Inventory for Men- International Index of Erectile Function (SHIM-IIEF) | At inclusion, 3 months, 6 months, 12 months and 24 months follow up.
  To evaluate other functional outcomes (sexual, hormonal and bowel functions) before and after FLA in men with prostate cancer by using validated questionnaires e.g. Sexual Health Inventory for Men- International Index of Erectile Function (SHIM-IIEF)
International Consultation on Incontinence Questionnaire (ICIQ) | At inclusion, 3 months, 6 months, 12 months and 24 months follow up.
  To evaluate other functional outcomes (sexual, hormonal and bowel functions) before and after FLA in men with prostate cancer by using validated questionnaires e.g. the International Consultation on Incontinence Questionnaire (ICIQ).
Quality of life using a validated quality of life questionnaire (EORTC QLQ PR25 | At inclusion , 3 months, 6 months, 12 months and 24 months follow up.
  To evaluate quality of life before and after FLA in men with prostate cancer by using a validated quality of life questionnaire (EORTC QLQ PR25).
Complication rate | At inclusion , 3 months, 6 months, 12 months and 24 months follow up.
  To evaluate the complication rate related to the technique

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen Fütterer, MD, PhD, Principal Investigator — Radboudumc Nijmegen; Michiel Sedelaar, MD, PhD, Principal Investigator — Radboudumc Nijmegen
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
The investigators will be author of submitted manuscripts in case they fulfill criteria for authorship according to regulations of scientific journals. After scientific publication of the results the study protocol, relevant data and findings will be made publically available for other centers to implement (parts) of this research into their standard clinical practice if they wish to do so.